CLINICAL TRIAL: NCT07001098
Title: Amino Acids for the Infant at Risk for Acute Kidney Injury After Cardiac Surgery: A Pilot Study
Brief Title: Amino Acids for Cardiac Surgery Associated AKI
Acronym: AKI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Shina Menon, Associate Professor, Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 80133
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury
Keywords: cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Amino Acids; amino-acid, glucose, and electrolyte solution; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amino acid (Experimental): Participants receive amino acids for up to 3 days starting at the time of their cardiac surgery
  Interventions: Drug: Amino Acids
- Placebo (Placebo Comparator): Participants receive equivalent volume of placebo for up to 3 days starting at the time of their cardiac surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amino Acids — The participants receive a continuous infusion of a balanced mixture of amino acids (Trophamine) in a dose of 2g/kg/day (max 100g/day) starting at the time of cardiac surgery up to 3 days
  Other Names: AA, Trophamine
  Arms: Amino acid
Drug: Placebo — The participants receive a continuous infusion of a lactated ringers (placebo), equivalent volume to amino acids, starting at the time of cardiac surgery up to 3 days
  Other Names: Lactated Ringer
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the feasibility of amino acid infusions in pediatric cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiac surgery and expected to be high risk

Exclusion Criteria:

* preoperative extracorporeal organ support
* CKD history (GFR<60ml/min/1.73m2 [≤1year] and GFR<90ml/min/1.73m2 [>1 year])
* serum creatinine defined preoperative AKI.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Amino acids Related Adverse Events | Baseline, Daily during infusion upto 48 hours after completion of infusion (upto 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Shina Menon, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No